CLINICAL TRIAL: NCT04499391
Title: COVID-19 Project ECHO for Nursing Homes: A Patient-centered, Randomized-controlled Trial to Implement Infection Control and Quality of Life Best Practice
Brief Title: COVID-19 Project ECHO in Nursing Homes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Jennifer Kraschnewski, Professor and Vice Chair for Research, Department of Medicine, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PCORI Nursing Homes
Record Dates: First submitted 2020-07-31; First posted 2020-08-05 (Actual); Results first posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Covid19
Keywords: Project ECHO; telehealth
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: stratified cluster randomized design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ECHO plus (Experimental): Nursing homes in this arm will receive the intervention via real-time, interactive videoconferencing using Zoom at no cost to participants. Sessions will be 90 minutes in duration and held weekly for 6 months (25 sessions total) at regularly scheduled times. Participants in this arm will receive a 2 month (8 sessions total) refresher course in Fall 2021. Project ECHO utilizes case-based, collaborative learning to support discussion of learners' challenges and barriers to guideline implementation
  Interventions: Other: Project ECHO
- ECHO (Active Comparator): Nursing homes in this arm will receive the intervention via real-time, interactive videoconferencing using Zoom at no cost to participants. Sessions will be 90 minutes in duration and held weekly for 6 months (25 sessions total) at regularly scheduled times. Project ECHO utilizes case-based, collaborative learning to support discussion of learners' challenges and barriers to guideline implementation
  Interventions: Other: Project ECHO

INTERVENTIONS:
Other: Project ECHO — Project ECHO utilizes case-based, collaborative learning to support discussion of learners' challenges and barriers to guideline implementation. This differentiates ECHO from traditional learning and facilitates rapid dissemination of medical knowledge and increased capacity to deliver best-practice care.studying innovative approaches.

SUMMARY:
Nursing homes are ground zero for the COVID-19 pandemic. Nursing homes are ill-equipped for the pandemic; though facilities are required to have infection control staff, only 3% have taken a basic infection control course. Significant research has focused on infection control in the acute care setting. However, little is known about the implementation of practices and effective interventions in long-term care facilities.The investigators propose an intervention utilizing Project ECHO, an evidence-based telehealth model, to connect Penn State University experts with remote nursing home staff and administrators to proactively support evidence-based infection control guideline implementation. Our study seeks to answer the critical research question of how evidence-based infection control guidelines can be implemented effectively in nursing homes

DETAILED DESCRIPTION:
The investigators will recruit 200 nursing homes with approximately 24,560 residents from across the United States through collaborations with our stakeholders. Nursing homes will be randomized to one of two arms: 1) AHRQ-funded COVID-19 ECHO that includes 16 weekly telehealth sessions addressing COVID-19 guidelines and best practices or 2) AHRQ-funded COVID-19 ECHO plus an additional 9 sessions with a focus on CDC infection control training. Randomization will be stratified by characteristics of nursing homes to ensure balance among the two trial groups, including size (number of beds),geographic location, and current COVID-19 infection rate. Patient-centered outcomes (nursing home residents with COVID-19 infections, hospitalizations, deaths, and QOL) will be assessed at baseline, 4, 6, 12, and 18 months. Our study is guided by the RE-AIM framework to critically evaluate both effectiveness and implementation outcomes of the proposed intervention. The RE-AIM framework is frequently utilized to improve sustainable adoption and implementation of effective, generalizable, evidence-based interventions like Project ECHO.

ELIGIBILITY:
Inclusion Criteria for Facilities Skilled Nursing Facility in United States Access to computer or electronic device

Exclusion Criteria for Facilities Previously participated in Project ECHO COVID-19 series either through Penn State or another institution

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2020-12-04 (Actual); Primary Completion 2022-09-27 (Actual); Study Completion 2022-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Kraschnewski, Principal Investigator — Penn State College of Medicine
Locations (1):
- Penn State College of Medicine, Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] D'Souza GC, Kraschnewski JL, Francis E, Heilbrunn E, Kong L, Lehman E, Osevala N, Urso J, Chamberlain L, Suda KM, McNeil L, Calo WA. Implementation of COVID-19 infection control best practices in nursing homes amid the pandemic. BMC Health Serv Res. 2024 Aug 17;24(1):941. doi: 10.1186/s12913-024-11407-z. PMID 39154191
- [Derived] Calo WA, Francis E, Kong L, Hogentogler R, Heilbrunn E, Fisher A, Hood N, Kraschnewski J. Implementing Infection Control and Quality of Life Best Practices in Nursing Homes With Project ECHO: Protocol for a Patient-Centered Randomized Controlled Trial. JMIR Res Protoc. 2022 May 13;11(5):e34480. doi: 10.2196/34480. PMID 35476823

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Nursing homes
Period: Overall Study
Arm/Group | ECHO Plus | ECHO
Started (Participants were not assigned to Arm/Groups) | NA; 68 Nursing homes (Participants were not assigned to Arm/Groups) | NA; 68 Nursing homes (Participants were not assigned to Arm/Groups)
Completed (Participants were not assigned to Arm/Groups) | NA; 64 Nursing homes (Participants were not assigned to Arm/Groups) | NA; 62 Nursing homes (Participants were not assigned to Arm/Groups)
Not Completed | NA; 4 Nursing homes | NA; 6 Nursing homes

BASELINE CHARACTERISTICS:
Population: Participants were not assigned to Arm/Groups and participant-level data were not collected.
  Participant age, gender and race/ethnicity data was not collected.
Units Other Than Participants: Nursing home
Groups:
- Total: Total of all reporting groups
Arm/Group | ECHO Plus | ECHO | Total
Number analyzed (Participants) | NA | NA | NA
Number analyzed (Nursing home) | 64 | 62 | 126
Age, Categorical [Count of Units; unit: Nursing home] — Participant age data was not collected. Population: Participant age data was not collected.
  Nursing home
    <=18 years | NA — Participants were not assigned to Arm/Groups and participant-level data were not collected | NA — Participants were not assigned to Arm/Groups and participant-level data were not collected | NA — Total not calculated because data are not available (NA) in one or more arms.
    Between 18 and 65 years | NA — Participants were not assigned to Arm/Groups and participant-level data were not collected | NA — Participants were not assigned to Arm/Groups and participant-level data were not collected | NA — Total not calculated because data are not available (NA) in one or more arms.
    >=65 years | NA — Participants were not assigned to Arm/Groups and participant-level data were not collected | NA — Participants were not assigned to Arm/Groups and participant-level data were not collected | NA — Total not calculated because data are not available (NA) in one or more arms.
Sex: Female, Male [Count of Units; unit: Nursing home] — Population: Participant gender was not collected.
  Nursing home
    Female | NA — Participants were not assigned to Arm/Groups and participant-level data were not collected | NA — Participants were not assigned to Arm/Groups and participant-level data were not collected | NA — Total not calculated because data are not available (NA) in one or more arms.
    Male | NA — Participants were not assigned to Arm/Groups and participant-level data were not collected | NA — Participants were not assigned to Arm/Groups and participant-level data were not collected | NA — Total not calculated because data are not available (NA) in one or more arms.
Race (NIH/OMB) [Count of Units; unit: Nursing home]
  American Indian or Alaska Native | NA — Participants were not assigned to Arm/Groups and participant-level data were not collected. | NA — Participants were not assigned to Arm/Groups and participant-level data were not collected. | NA — Total not calculated because data are not available (NA) in one or more arms.
  Asian | NA — Participants were not assigned to Arm/Groups and participant-level data were not collected. | NA — Participants were not assigned to Arm/Groups and participant-level data were not collected. | NA — Total not calculated because data are not available (NA) in one or more arms.
  Native Hawaiian or Other Pacific Islander | NA — Participants were not assigned to Arm/Groups and participant-level data were not collected. | NA — Participants were not assigned to Arm/Groups and participant-level data were not collected. | NA — Total not calculated because data are not available (NA) in one or more arms.
  Black or African American | NA — Participants were not assigned to Arm/Groups and participant-level data were not collected. | NA — Participants were not assigned to Arm/Groups and participant-level data were not collected. | NA — Total not calculated because data are not available (NA) in one or more arms.
  White | NA — Participants were not assigned to Arm/Groups and participant-level data were not collected. | NA — Participants were not assigned to Arm/Groups and participant-level data were not collected. | NA — Total not calculated because data are not available (NA) in one or more arms.
  More than one race | NA — Participants were not assigned to Arm/Groups and participant-level data were not collected. | NA — Participants were not assigned to Arm/Groups and participant-level data were not collected. | NA — Total not calculated because data are not available (NA) in one or more arms.
  Unknown or Not Reported | NA — Participants were not assigned to Arm/Groups and participant-level data were not collected. | NA — Participants were not assigned to Arm/Groups and participant-level data were not collected. | NA — Total not calculated because data are not available (NA) in one or more arms.
Location [Count of Units; unit: Nursing home] — Rural/urban
  Nursing home
    Rural | 26 | 27 | 53
    Urban | 38 | 35 | 73
Facility Size [Count of Units; unit: Nursing home]
  <60 Beds | 17 | 19 | 36
  >=60 beds | 47 | 43 | 90
Facility Payment Model [Count of Units; unit: Nursing home]
  For-profit | 41 | 33 | 74
  Not-for-profit | 23 | 29 | 52
Facility Type [Count of Units; unit: Nursing home]
  Independent | 27 | 32 | 59
  Networked | 37 | 30 | 67
Memory Care Status [Count of Units; unit: Nursing home]
  Yes | 17 | 10 | 27
  No | 47 | 52 | 99
Baseline Infection Rate [Count of Units; unit: Nursing home] — Some vs. none
  Nursing home
    Some | 53 | 55 | 108
    None | 11 | 7 | 18

OUTCOME MEASURES:

1. Primary Outcome: Infection Rate
Description: Rate of COVID-19 infection in enrolled nursing homes, as measured by the cumulative 4-week incidence at study points for Confirmed COVID-19 cases per 1,000 residents
Time Frame: Baseline, 4, 6, 12, 18 months
Population: Nursing homes were assigned to Arms/Groups, participant level data is not available
Measure: Mean (Standard Deviation); unit: infections per 1,000 residents in 4 week
Units Other Than Participants: Nursing home
Arm/Group | ECHO Plus | ECHO
Number analyzed (Participants) | NA | NA
Number analyzed (Nursing home) | 64 | 64
infections per 1,000 residents in 4 week
  Baseline | 141.91 (266.23) | 106.57 (192.49)
  4m | 1.54 (6.62) | 2.86 (14.11)
  6m | 2.08 (16.67) | 0.83 (5.04)
  12m | 28.01 (54.48) | 26.56 (50.17)
  18m | 33.07 (66.81) | 30.5 (74.18)

2. Secondary Outcome: Hospitalization
Description: Number of COVID-19 hospitalizations from enrolled nursing homes, as measured by Cumulative 4-week incidence at study points for Total COVID-19 admissions
Time Frame: Baseline, 4, 6, 12, 18 months
Population: Nursing homes were assigned to Arms/Groups, participant level data is not available
Measure: Mean (Standard Deviation); unit: per 1,000 residents in 4 weeks
Units Other Than Participants: Nursing home
Arm/Group | ECHO Plus | ECHO
Number analyzed (Participants) | NA | NA
Number analyzed (Nursing home) | 64 | 62
per 1,000 residents in 4 weeks
  Baseline | 40.05 (83.13) | 39.12 (83.88)
  4m | 3.09 (14.01) | 4.72 (21.33)
  6m | 5.55 (30.40) | 5.18 (37.47)
  12m | 24.57 (113.55) | 7.87 (24.71)
  18m | 7.27 (21.31) | 13.58 (55.54)

3. Secondary Outcome: Death
Description: Number of COVID-19 deaths from enrolled nursing homes, as measured by Cumulative 4-week incidence at study points for Total COVID-19 deaths
Time Frame: Baseline, 4, 6, 12, 18 months
Population: Nursing homes were assigned to Arms/Groups, participant level data is not available
Measure: Mean (Standard Deviation); unit: per 1,000 residents in 4 weeks
Units Other Than Participants: Nursing home
Arm/Group | ECHO Plus | ECHO
Number analyzed (Participants) | NA | NA
Number analyzed (Nursing home) | 64 | 62
per 1,000 residents in 4 weeks
  Baseline | 30.22 (61.59) | 31.98 (66.2)
  4m | 0.82 (4.39) | 0.00 (0.00)
  6m | 0.46 (2.61) | 0.30 (2.35)
  12m | 3.60 (12.51) | 3.71 (11.37)
  18m | 2.00 (7.28) | 0.19 (1.49)

4. Secondary Outcome: Flu-like Illness
Description: Number of flu-like illnesses reported from enrolled nursing homes, as measured by Cumulative 4-week incidence at study points for Total confirmed new influenza per 1,000 residents in 4 weeks
Time Frame: Baseline, 4, 6, 12, 18 months
Population: Nursing homes were assigned to Arms/Groups, participant level data is not available
Measure: Mean (Standard Deviation); unit: per 1,000 residents in 4 weeks
Units Other Than Participants: Nursing home
Arm/Group | ECHO Plus | ECHO
Number analyzed (Participants) | NA | NA
Number analyzed (Nursing home) | 64 | 62
per 1,000 residents in 4 weeks
  Baseline | 0.65 (5.21) | 0.00 (0.00)
  4m | 0.00 (0.00) | 0.00 (0.00)
  6m | 0.00 (0.00) | 0.62 (4.88)
  12m | 0.35 (2.78) | 1.36 (8.01)
  18m | 0.00 (0.00) | 0.00 (0.00)

ADVERSE EVENTS:
Time Frame: Adverse event data were not collected as patients were not enrolled in the study. This study included only secondary data.
Description: Adverse event data were not collected as patients were not enrolled in the study. This study included only secondary data.
Arm/Group | ECHO Plus | ECHO
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-12): https://cdn.clinicaltrials.gov/large-docs/91/NCT04499391/Prot_SAP_000.pdf